CLINICAL TRIAL: NCT02288702
Title: Comparison of Bispectral Index Values in Patients With and Without Down's Syndrome
Status: Terminated | Type: Observational
Why Stopped: lack of recruitment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Priti G. Dalal, Associate Professor, Milton S. Hershey Medical Center
Other Study IDs: STUDY00000604
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: This is the group with no neurological problems or syndrome
  Interventions: Device: monitoring BIS in both groups
- Down syndrome: This is the group with Down syndrome
  Interventions: Device: monitoring BIS in both groups

INTERVENTIONS:
Device: monitoring BIS in both groups — We will be monitoring BIS in both groups. A BIS monitor may be placed prior to induction or immmeditaely afterwards for monitoring BIS. All patients will receive general anesthesia. A standard inhalation induction agent such as sevoflurane and oxygen will be administered via face mask with or without an oral airway. An inhalation agent will be administered for the duration of the procedure. The MAC goal for inhalation agents will be 1. If the patient moves, the MAC goal will be increased to 1.5 and this change will be recorded.
  Other Names: BIS

SUMMARY:
About 1 in every 700 babies born in the United States has Down's Syndrome (DS; Trisomy 21), 99% of whom have some degree of intellectual disability. Recent advances in medicine have resulted in a dramatically improved lifespan of about 25 to 60 years of age. Yet, there is limited data about anesthetic management in this increasing patient population. The bispectral index (BIS) monitor is a non-invasive monitoring device that reports a value between 0 and 100correlating to level of consciousness of an individual. A value of 0 indicates lack of brain activity while 100 indicates an awake/alert state. This monitor can be used to assess the depth of anesthesia. Patients with intellectual disability from congenital neurological diseases have lower BIS values compared to patients without any neurological impairment (Valkenburg 2009). The results may suggest that DS patients would require less anesthetic drugs compared to patients without any neurological impairment. To date, there are no studies in DS patients.

DETAILED DESCRIPTION:
Based on the Valkenburg group's study (2009), one might hypothesize that if the BIS value is fixed for all patients, then a patient with an intellectual disability such as a patient with DS would require less anesthetic drugs compared to a control patient without any neurological disability. However, if one is only using a clinical sedation scale, the DS patient may receive more anesthetic drugs in order to achieve the same level of clinical unconsciousness as a patient without DS.

This project seeks to elucidate the effect of anesthetic techniques and agents on patients with DS compared to those without DS and any intellectual disability. The goal of this project is to compare BIS values in patients with DS to those without DS undergoing a standardized general anesthetic technique. The investigators hypothesize that patients with DS would have lower (>25%) BIS values compared to those without DS.

Known potential sources of artifact signals that could change BIS values include electromyographic activity, electric devices, hypothermia, hypoglycemia, and the timing and type of anesthetics used (Duarte 2009, Dahaba 2005). These potential sources will be identified and reported during the study, and those patients will be excluded from the study

ELIGIBILITY:
Inclusion Criteria:

* • Patients with DS and those without DS receiving BIS monitoring

  * Children between the ages of 2 and 17 years old (inclusive)
  * Patients scheduled for unilateral or bilateral tympanostomy (ear tube placement) at Penn State Hershey Medical Center
  * Patients with American Society of Anesthesiologists (ASA) physical status I, II and III
  * Eligible for standard general anesthesia technique protocol as determined by anesthesia provider(s)

Exclusion Criteria:

* Patients with congenital diseases/anomalies except Down's Syndrome
* Patients with myotonic dystrophies or other neurodegenerative diseases
* Patients with cerebrovascular accidents (strokes)
* Patients not receiving BIS monitoring
* Pregnant patients
* Patients with allergic skin reactions to electrode patches
* Patients 18 years of age and greater

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 2-17 years (inclusive) scheduled for tympanostomy on the 24-hr and 48-hr operating room (OR) schedules
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

PRIMARY OUTCOMES:
measure BIS values in the normal patients and those with Down syndrome under anesthesia | 2 years
  >25% lower BIS values in patients with DS compared to patients without DS

CONTACTS AND LOCATIONS:
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States